CLINICAL TRIAL: NCT04630886
Title: Local Injection of Tranexamic Acid May Reduce Bleeding, Injection Pain, and Other Post-op Complications During Mohs Micrographic Surgery
Brief Title: Use of Tranexamic Acid in Reduction of Post-Op Complications in Mohs Micrographic Surgery
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Drug supply issues
Sponsor: Riley McLean (Other)
Responsible Party: Sponsor-Investigator, Riley McLean, Principle Investigator, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H00019337
Record Dates: First submitted 2020-11-02; First posted 2020-11-16 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Skin Neoplasms
MeSH Terms: conditions — Skin Neoplasms | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Once a participant has provided informed consent to participate in the study, he/she will be randomly assigned to either the TXA experimental group or the control group. A randomized list will be created prior to the start of the study with the help of a biostatistician. The provider will be aware of which study arm the participant is in, however the participant will be blinded.
Who Masked: Participant
Masking Description: The surgeon performing the Mohs surgery will be aware of which group the participant is in. The participant will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tranexamic acid (Experimental): The TXA group will receive 2% lidocaine with 1:100,000 epinephrine mixed 50/50 with 50mg/ml TXA (with 50% dilution, this will yield 1% lidocaine with 1:200,000 epi).
  Interventions: Drug: Tranexamic acid injection; Drug: Lidocaine Epinephrine
- Control (Active Comparator): The control group will use the routine local anesthetic of buffered 1% lidocaine with 1:200,000 epinephrine.
  Interventions: Drug: Lidocaine Epinephrine

INTERVENTIONS:
Drug: Tranexamic acid injection — subcutaneous injection of 50mg/ml TXA
  Arms: Tranexamic acid
Drug: Lidocaine Epinephrine — subcutaneous injection of 1% lidocaine mixed with 1:200,000 epinephrine

SUMMARY:
The purpose of this study is to evaluate the use of locally injected tranexamic acid (TXA) under the skin during Mohs micrographic surgery for removal of skin cancers in patients on anticoagulation. TXA may be helpful in reducing bleeding and pain during surgery, and may also lead to fewer post-operative complications following surgery such as graft loss, specifically in patients on blood-thinners.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the efficacy of subcutaneous infiltration of tranexamic acid (TXA) in the reduction of peri- and post-operative complications including bleeding, infections, flap and graft loss in anticoagulated patients undergoing Mohs micrographic surgery. A secondary objective is to evaluate the ability of TXA to increase the pH of lidocaine with epinephrine, and whether it causes less pain than the alternative during injection of local anesthetic.

TXA may serve as an effective local antifibrinolytic agent to decrease perioperative and postoperative bleeding while also causing less injection pain in patients undergoing Mohs surgery.

Background:

TXA is a well-established antifibrinolytic agent used in many surgical fields to effectively reduce post-operative bleeding. TXA is a synthetic lysine analogue that prevents the lysis of polymerized fibrin in blood clots. It has been used intravenously, orally, and subcutaneously to reduce bleeding during orthopedic procedures, to manage postpartum bleeding, and in trauma patients to control significant hemorrhage. It has also been used intravenously to reduce the need for blood transfusions in cardiac and liver transplantation.The safety of TXA has been verified in numerous publications across multiple medical specialties. Additionally, the pH of TXA ranges from 6-8, indicating that it may serve as an effective buffering agent and cause less pain with injection of anesthetic agents.

Many institutions have begun to use tranexamic acid to reduce postoperative bleeding. The medication is now readily available in the Pyxis of the investigators. The use of TXA within the wound bed and underlying undermined edges of flaps performed in patients who are anticoagulated is becoming the standard of care. Anecdotally, this has been quite successful in reducing post operative bruising and post operative bleeding requiring an emergency visit. In this protocol, the study arm involving the use of TXA and the study arm without the use of TXA are currently standard of care and are currently routinely used intraoperatively in clinical practice.

The investigators are performing this study to examine the efficacy of TXA as a safe, local antifibrinolytic agent in dermatologic surgeries and will analyze postoperative bleeding as well as other postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Must be on systemic anticoagulation therapy (indirect or direct anticoagulants or anti-platelet agents)
* Must be scheduled for Mohs surgery at the University of Massachusetts Department of Dermatology

Exclusion Criteria:

* History of hypercoaguable disorder (e.g. Factor V Leiden Deficiency)
* History of deep vein thrombosis or pulmonary embolism
* Systolic blood pressure greater than 200 on day of surgery
* Known allergy to TXA
* Currently taking systemic retinoids
* Unable to consent
* Pregnant women
* Prisoners

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2024-01-16 (Actual)

PRIMARY OUTCOMES:
Postoperative Complications | From day of surgery to 12 weeks post-operation
  Primary outcome measures will be the number of postoperative complications, including infection, bleeding (necessitating phone calls to providers or additional clinic visits), hematoma formation, and flap or graft failure.

SECONDARY OUTCOMES:
Hemostasis | during surgery
  The quality of intraoperative hemostasis will be measured on a 1-4 scale titled "Quality of the Field", with 1 being "excellent, better than expected/predicted for this procedure" and 4 being "poor, oozing that required adding gauze dressing and local pressure" (the higher the score, the worse the outcome)
Injection Pain | 30 minutes post initial injection
  Injection pain will be measured via self reported pain intensity within the first 30 minutes of initial injection on the day of surgery. The pain scale is scored 0-10 (0 = no pain; 10 = unable to move). The higher the score, the worse the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Riley McLean, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zilinsky I, Barazani TB, Visentin D, Ahuja K, Martinowitz U, Haik J. Subcutaneous Injection of Tranexamic Acid to Reduce Bleeding During Dermatologic Surgery: A Double-Blind, Placebo-Controlled, Randomized Clinical Trial. Dermatol Surg. 2019 Jun;45(6):759-767. doi: 10.1097/DSS.0000000000001786. PMID 30640775
- [Background] Poeran J, Rasul R, Suzuki S, Danninger T, Mazumdar M, Opperer M, Boettner F, Memtsoudis SG. Tranexamic acid use and postoperative outcomes in patients undergoing total hip or knee arthroplasty in the United States: retrospective analysis of effectiveness and safety. BMJ. 2014 Aug 12;349:g4829. doi: 10.1136/bmj.g4829. PMID 25116268